CLINICAL TRIAL: NCT06031610
Title: Revascularization Effect on CSVD Burden in Carotid Artery Stenosis
Acronym: RECAS
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZJPPHEC2023O（290）
Record Dates: First submitted 2023-08-21; First posted 2023-09-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-10

CONDITIONS: Carotid Artery Stenosis; Cerebral Small Vessel Diseases
Keywords: Carotid Artery Stenosis; Cerebral Small Vessel Diseases; Revascularization; Carotid artery stenting; prospective cohort
MeSH Terms: conditions — Carotid Stenosis; Cerebral Small Vessel Diseases | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals accepted CAS: Procedure: CAS and Standard medical treatment.
  Other:
  1. Neuropsychological testing.
  2. Multimodal CT: included NCCT+CTP and reconstructed 4D-CTA.
  3. Multimodal MRI included T1, T2-FLAIR, DWI, DTI, SWI, fMRI.
  4. Optical coherence tomography angiography.
  Interventions: Procedure: carotid artery stenting; Drug: drug therapy
- Individuals accepted standard medical treatment alone.: Procedure: Standard medical treatment alone.
  Other:
  1. Neuropsychological testing.
  2. Multimodal CT: included NCCT+CTP and reconstructed 4D-CTA.
  3. Multimodal MRI includedT1, FLAIR, MRA, PWI and/or ASL, DTI, DKI, SWI, fMRI.
  4. Optical coherence tomography angiography.
  Interventions: Drug: drug therapy

INTERVENTIONS:
Procedure: carotid artery stenting — Patients were monitored for at least 24 h after surgery, with control for hyperperfusion syndrome, dual antiplatelet therapy was continued for 4-6 weeks, and the postoperative patients have the final residual stenosis of less than 30%, thrombolysis in Myocardial Infarction (TIMI) grade 3, and no dissection or thrombosis. Any surgery-related complications were recorded.
  Groups: Individuals accepted CAS
Drug: drug therapy — Carotid artery stenosis requires taking antiplatelet aggregation drugs and statin lipid-lowering drugs. It can inhibit platelet aggregation, stabilize plaque, reduce vascular inflammatory factors, and prevent further development of atherosclerosis.

SUMMARY:
RECAS is a prospective cohort of 1,000 patients with carotid artery stenosis (CAS) and undergoing revascularization therapy or standard medication treatment alone. The goal of this study is to validate whether CAS revascularization when compared to standard medication treatment alone, can effectively reduce the progression of Cerebral small vessel disease (CSVD) burden, as well as improve the severity of retinal pathologies and cognitive impairment. Therefore, Patients aged ≥ 40 years have more than 50% stenosis in unilateral carotid artery and sign informed consent will be recruited. In this study, patients will be asked to undergo Computed Tomography Angiography (CTA)/ Digital Subtraction Angiography (DSA), Computed Tomography Perfusion (CTP),multimodal Magnetic Resonance Imaging (MRI), Optical Coherence Tomography Angiography (OCTA) and neuropsychological testing. Estimated follow-up can be up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 40 years.
2. ≥ 50% stenosis in unilateral carotid artery.
3. Sign informed consent.

Exclusion Criteria:

1. Previous history of major head trauma and any intracranial surgery
2. Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage, and other space occupying lesions
3. Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement.
4. Severe loss of vision, hearing, or communicative ability.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population for this study consists of patients who have been diagnosed with Carotid Artery Stenosis. The inclusion criteria are: Patients aged ≥ 40 years，≥ 50% stenosis in unilateral carotid artery,sign informed consent.The exclusion criteria are: Previous history of major head trauma and any intracranial surgery,intracranial abnormalities,extrapyramidal symptoms or mental illness which may affect neuropsychological measurement,severe loss of vision, hearing, or communicative ability. The patients will be recruited from Zhejiang Provincial People's Hospital in the city of Hangzhou.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
The development of total brain small vessel disease burden in MRI | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Total brain small-vessel disease burden is used to assess the overall impact of CSVD, with a score range of 0-4 points.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  To assess changes in cognitive function of patients.
Mini-mental State Examination(MMSE) score | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  To assess changes in cognitive function of patients.
Blood flow density | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Record blood flow density (%) of OCTA.
Vascular perfusion area | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Record vascular perfusion area (mm^2) of OCTA.
Macular fovea retinal thickness | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Record macular fovea retinal thickness (μm) of OCTA.
Retinal nerve fiber layer thickness | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Record retinal nerve fiber layer thickness (μm) of OCTA.
Change of the volume of hypoperfusion (delay time>3s from baseline to follow-up CTP). | baseline,3-month,6-month, and every 1 year, follow-up time up to 10 years.
  Change of the volume of delay time>3s in follow-up minus the volume at baseline.
Stenosis percent | baseline,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Restenosis can be identified by CTA/DSA evaluating the percentage of lumen of vessel but can also be classified as symptomatic vs asymptomatic and/or requiring or not re-intervention.
Number of Patients with cerebrovascular events, cardiovascular events or death | baseline,1-month,3-month,6-month,and every 1 year, follow-up time up to 10 years.
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage and cerebral hyperperfusion syndrome. Cardiovascular events included angina and myocardial infarction. Death included any reason caused death.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duering M, Biessels GJ, Brodtmann A, Chen C, Cordonnier C, de Leeuw FE, Debette S, Frayne R, Jouvent E, Rost NS, Ter Telgte A, Al-Shahi Salman R, Backes WH, Bae HJ, Brown R, Chabriat H, De Luca A, deCarli C, Dewenter A, Doubal FN, Ewers M, Field TS, Ganesh A, Greenberg S, Helmer KG, Hilal S, Jochems ACC, Jokinen H, Kuijf H, Lam BYK, Lebenberg J, MacIntosh BJ, Maillard P, Mok VCT, Pantoni L, Rudilosso S, Satizabal CL, Schirmer MD, Schmidt R, Smith C, Staals J, Thrippleton MJ, van Veluw SJ, Vemuri P, Wang Y, Werring D, Zedde M, Akinyemi RO, Del Brutto OH, Markus HS, Zhu YC, Smith EE, Dichgans M, Wardlaw JM. Neuroimaging standards for research into small vessel disease-advances since 2013. Lancet Neurol. 2023 Jul;22(7):602-618. doi: 10.1016/S1474-4422(23)00131-X. Epub 2023 May 23. PMID 37236211
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37236211/